CLINICAL TRIAL: NCT04909762
Title: Feasibility of Implementing the Paediatric Early Rehabilitation & Mobilisation During InTensive Care (PERMIT) Intervention
Brief Title: Paediatric Early Rehabilitation & Mobilisation During InTensive Care (PERMIT) Feasibility
Acronym: PERMIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Birmingham (Other)
Collaborators: King's College Hospital NHS Trust (Other); University Hospital Southampton NHS Foundation Trust (Other); Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERN_18-1134
Record Dates: First submitted 2021-05-11; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-03

CONDITIONS: ICU; Critical Illness
Keywords: PICU; Paediatric; Early mobilisation; Early rehabilitation; Observational
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: All patients will receive Early Rehabilitation and Mobilisation intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early rehabilitation and mobilisation (Other): Early rehabilitation/mobilisation (ERM) encompasses patient-tailored interventions, delivered individually or in a bundled package, provided by health care professionals from multiple disciplines and parents/carers within intensive care settings to promote recovery, both physical (e.g. movement, functional activities, ambulation) and non-physical (e.g. speech, play, psychological, cognitive). In adult intensive care, ERM has been shown in clinical trials to improve long term physical functioning and return to independence. It can also shorten the length of ventilation and stay in intensive care and hospital with significant economic benefit.
  Interventions: Other: Early Rehabilitation and Mobilisation (ERM)

INTERVENTIONS:
Other: Early Rehabilitation and Mobilisation (ERM) — Early rehabilitation/mobilisation (ERM) encompasses patient-tailored interventions, delivered individually or in a bundled package. It is provided by health professionals from multiple disciplines and care-givers within intensive care settings.

SUMMARY:
19,000 children and young people (CYP)/year are admitted to Paediatric Intensive Care Unit (PICU). The investgators want to see if patients recover quicker if rehabilitation starts early and they are encouraged to get moving whilst still in PICU. This is known as 'early rehabilitation and mobilisation' (ERM).

PERMIT is an National Institute of Health research/Health Technology Assessment funded programme with four stages:

1. The investgators undertook a national survey of perceptions, a systematic review of the literature and an observational study of ERM over 2 weeks across 14 United Kingdom PICUs
2. The investgators worked with professionals and families to develop an ERM manual appropriate for the age and acuity level of the child.
3. In the current phase the investgators will try out the ERM manual in 3 PICUs to see if they are useful and then
4. Make suggestions about further research.

This protocol outlines the third stage, exploring feasibility and acceptability of implementing the PERMIT intervention in the following Steps:

Step 1: Implementing the PERMIT intervention within 3 PICUs Step 2: Enrolling and delivering PERMIT intervention to CYP in PICU Step 3: Measuring outcomes and assessing impact of PERMIT intervention on CYP and parents.

Over 5 months, the investgatorswill share the ERM manual with 6-15 key staff on 3 PICUs so that they can consider implementation; they will be interviewed weekly. 90 staff will be eligible to complete 3 online questionnaires. If implementation is feasible, the investgators will recruit up 30 children aged 0-16 years in 3 PICUs if parents consent. On ward rounds the PICU team will use the ERM manual to assess acuity and prescribe ERM. the investgators will collect routine data and observe whether prescribed ERM is delivered. After further consent, up to 30 parents can complete questionnaires at PICU discharge and interviews (n=12-15 consenting, approx 3 declining Step 2) within 30 days. 12-15 staff will be interviewed.

DETAILED DESCRIPTION:
Purpose and design To design clinical trials to investigate the potential benefits of ERM in critically ill children, it is crucial to understand the feasibility of implementation and opinions of families.

The Stage 3 feasibility study aims to assess the feasibility of the following Steps:

Step 1:

(i) Prepare PICUs to implement the PERMIT intervention. (ii) Assess barriers & facilitators to implementation.

Step 2:

(iii) Assess enrolment, recruitment and delivery of the PERMIT intervention to CYP.

(iv) Monitor safety of the PERMIT intervention and related adverse events.

Step 3:

(v) Measure clinically important outcomes following delivery of the PERMIT intervention.

(vi) Assess parent/legal guardian acceptability of the PERMIT intervention and future trial design.

Recruitment Recruitment for the PERMIT Stage 3 feasibility study will take place on 3 PICUs in United Kingdom National Health Service Trusts: Birmingham's Children's, University hospital Southampton, and King's College hospital In Steps 1-3, the investgators will recruit Health care practitioners and managers within PICU For Steps 2-3 the investgators will recruit Children and Young People (CYP) For Step 3 the investgators will recruit Parents/legal guardians and CYP fulfilling criteria above Screening, recruitment and consent All screening, recruitment and consent will be managed by the Local and Central PERMIT Research Teams: Local PERMIT Research Team: Each of the three participating PICU sites will identify a Principal Investigator, supported by a therapist/nurse. This will form the Local PERMIT Research Team, who will provide local data collection at the sites.

Central PERMIT Research Team: The Chief Investigator and the PERMIT Trial Management Group will form the Central PERMIT Research Team and provide support, oversight and centralised data collection across the sites. The investgators require agreement and consent at a PICU level to prepare the PICU for implementing the PERMIT intervention (step 1) and to deliver the PERMIT intervention to CYP (step 2). PICU-level consent will be provided by the Clinical Lead during the local R&D trial approval process for the PERMIT feasibility study. This provides consent for the unit to engage in implementing the PERMIT intervention and follow the specified implementation process in the PERMIT intervention manual.

PICU-level approval will also provide permission for the Local PERMIT Research Team to approach PERMIT champions for the weekly debrief and PICU health care professionals for the three brief online surveys, as described below.

Step 1:

Step 1 will assess the feasibility of implementing the preparation phases of the PERMIT intervention in the three PICUs (i.e. phase 1 'build the team', phase 2 'take stock', phase 3 'get buy-in' and phase 4 'get ready').

PERMIT champions: Following Research Ethics Committee and local R&D approval, the Local PERMIT Research Team at each site will share the protocol and the PERMIT intervention manual with the medical, nursing and therapy leads within their PICU to nominate and 'build the team' of PERMIT champions. The Local PERMIT Research Team will provide the PERMIT champions with an email invitation, participant information sheet, and consent form regarding taking part in the weekly debrief. Consent forms will be completed with a member of the Local PERMIT research team.

PICU health care professionals: The Local PERMIT Research Team at each site will use internal email lists to invite all multidisciplinary PICU health care professionals to complete the first brief online survey. They will send an email invitation after the health care professionals have received education about the PERMIT intervention from the PERMIT champions, but before any patient recruitment starts. The email invitation will have a participant information sheet attached. Both these documents highlight that completion and submission of the survey is an indicator of informed consent. Therefore, no separate consent form will be required.

Completed surveys are automatically submitted via web-based survey tool (SmartSurvey) to the Central PERMIT Research Team for processing and analysis. The Central PERMIT Research Team will monitor survey responses to ensure that relevant health care professional groups and the three PICUs are represented. If required, the Local PERMIT Research Team at each site will send the email invitation again to specific under-represented groups. This will ensure that the investgators have representatives from all three units, from different health care professional groups and from people who have had a variety of experiences.

Step 2:

After phases 1-4 have been implemented, study sites will progress to step 2 which will assess the feasibility of implementing the delivery phases of the PERMIT intervention (i.e. phase 5 'make it work' and phase 6 'keep it going').

PERMIT champions: The weekly debrief with PERMIT champions will continue. PICU health care professionals: The Local PERMIT Research Team at each site will invite all multidisciplinary PICU health care professionals to complete the second brief online survey, following the same process as described for step 1.

CYP: The investgators will display a poster about the PERMIT feasibility study in public areas in each PICU. Basic information about the study, in the form of an awareness leaflet, will be provided to all parents/legal guardians of CYP admitted to PICU during the study period.

In conjunction with patient's clinical team, the local PERMIT Research Team will screen and recruit CYP to receive the PERMIT intervention. They will screen all CYP admitted to each PICU against the study inclusion and exclusion criteria and record the screening and all related decisions in the screening log at each site. They will approach the parents/legal guardians of eligible CYP on day 1 or 2 of admission (where possible). They will explain the study and provide the participant information sheet.

After providing time for parents/legal guardians to read the information and consider the study, the Local PERMIT Research Team will return to ask for consent for the CYP to take part in the study using the consent form. They will discuss the different options for consent. At this point, parents/legal guardians can choose between the following:

Consenting for CYP to receive the PERMIT intervention, with accompanying data collection (specifically, CYP clinical data, PERMIT intervention data and safety monitoring). No additional requirements for parents/legal guardians.

If they consent to the PERMIT intervention, they can also consent to complete additional outcome measurement tools (e.g. related to quality of life, fatigue, pain).

If they consent to the PERMIT intervention and complete additional outcome measurement tools, they can also consent to an optional interview to assess acceptability.

Consent from parents/legal guardians will be obtained by a member of the Local PERMIT Research Team, with copies provided to the parents/ legal guardians and for the medical notes.

The majority of CYP will be unable to provide assent to participate (for example; because of their age (<1 year of age), on pain relief medications, sedated to tolerate interventions). Therefore, the investgators will rely primarily on consent from parents/legal guardians. However, where possible and appropriate, the Local PERMIT Research Team will seek verbal or written assent from the CYP themselves, where consent has first been obtained from their parent/legal guardian. Assent will be recorded on a CYP assent form, which will be completed with a member of the Local PERMIT Research Team with copies provided to parents/legal guardians and for the medical notes.

During the assenting process, the Local PERMIT Research Team will ensure that CYP:

* Understand the purpose and nature of the research.
* Understand what the research involves, its benefits, risks and burdens.
* Understand the alternatives to taking part.
* Are able to retain the information long enough to make an effective decision.
* Are able to make a free choice.
* Are capable of making this particular decision at the time it needs to be made (recognising that their capacity may fluctuate, and they may be capable of making some decisions but not others depending on their complexity).

The Local PERMIT Research Team will employ a 'best interests' approach. Mental capacity will be assumed unless proven otherwise. All members of the Local PERMIT Research Team recruiting CYP into this study will have been trained in Mental Capacity Assessment as part of routine clinical training.

Parents/legal guardians and CYP may request withdrawal from the PERMIT feasibility study at any point, including during step 2 where they have agreed for their child to receive the PERMIT intervention. Reasons for withdrawal will be recorded in the screening logs at each PICU site. At the time of withdrawal the investgators will ascertain if they wish to withdraw from ongoing involvement in the PERMIT intervention or if they wish for all their previously collected data to be removed.

Step 3:

PERMIT champions: The weekly debrief with consenting PERMIT champions will continue.

PICU health care professionals: The Local PERMIT Research Team at each site will invite all multidisciplinary PICU health care professionals to complete the third and final brief online survey, following the same process as described for steps 1-2.

At the end of each of the three brief online surveys, health care professionals will be asked if they would be willing to consider taking part in an interview. If they indicate yes, they will be asked to provide their name and email address. Their name and email address will not be linked to any of their survey responses. Completed surveys - and any names and email addresses provided - are automatically submitted to the Central PERMIT Research Team for processing and analysis.

To recruit health care professionals for the interviews, the investgators will use two approaches: (i) the Central PERMIT Research Team will send an email invitation to survey respondents who agreed to consider taking part in an interview, and (ii) the Local PERMIT Research Team will send the same email invitation asking for participants from specific under-represented groups or groups that the investgators are particularly keen to hear from. This two-pronged approach will ensure that the investgators have representatives in the interviews from all three units, from different health care professional groups and from people who have had a variety of experiences of the PERMIT intervention.

The Participant Information Sheet and consent form will be sent by email to the potential participant by the researcher from the Central PERMIT Research Team. Participants will be asked to complete and return the consent form via email to a secure nhs.net address. Prior to commencing the interview the participant information sheet will be discussed and consent re-affirmed verbally.

Health care professionals responses to the on line survey cannot be withdrawn as they are anonymous. Health care professionals may withdraw their consent to participate during or after an interview. The investgators will ask permission to use any information already provided. If participants do not provide this permission, the investgators will remove all data.

CYP: Throughout step 3, the Local PERMIT Research Team will continue to screen and recruit CYP to receive the PERMIT intervention, as described in step 2.

Parents/legal guardians of CYP receiving the PERMIT intervention: The Local PERMIT Research Team will re- approach parents/legal guardians of the CYP included in step 2 who also agreed to complete additional outcome measurement tools (e.g. related to quality of life, fatigue, pain) and may also have agreed to take part in an interview to assess acceptability.

The Local PERMIT Research Team will re-approach parents/legal guardians of the CYP included in step 2 who only agreed only for their child to receive the PERMIT intervention with accompanying data collection.

ELIGIBILITY:
Inclusion Criteria:

* Steps 1-3:

The PERMIT champions: health care professionals (HCP) and managers from each PICU who will lead the implementation of the PERMIT intervention. The PERMIT champions could be the PI, the PIC manager, a consultant lead, a physio lead and a senior nurse but this is decided locally.

HCP: Health care professionals who work within the PICU and could be /are involved in delivering the PERMIT intervention to CYP (i.e. doctors, nurses, allied health professionals, play therapists, psychologists etc.).

• Steps 2-3:

CYP

Inclusion:

Admitted to a participating PICU. Age 0 to <16 years at time of admission. Likely to remain within PICU on day 3 post admission. Consent by parent/legal guardian.

• Step 3:

Parents/legal guardians of CYP fulfilling criteria above.

Exclusion Criteria:

• Steps 1-3:

PERMIT champions who decline to participate in the debrief.

• Steps 2-3:

Local decision by PICU health care professionals not to include CYP.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Number of PICUs implementing PERMIT intervention | 4 weeks
  The prevalence and scope of ERM will be described as the proportion of PICUs progressing from step 1 (PICU preparation) to step 2 (patient delivery).
  Assessment of implementation progress within PICUs (e.g. barriers and facilitators to implementation) PICUs using the weekly debrief with PERMIT champions, the three brief online surveys of PICU health care professionals and the interviews with PICU health care professionals.
Proportion of eligible CYP recruited to receive the PERMIT intervention | 4 weeks
  The proportion of eligible CYP recruited to receive the PEMRIT intervention will be calculated as the number of eligible CYP recruited divided by the total number of eligible CYP at each site.
Proportion of completed outcome assessment tools of eligible CYP | 4 weeks
  Proportion of CYP with 100% completed outcome measurement tools and >50% completed will be recorded at each PICU site.

SECONDARY OUTCOMES:
Acceptability of all data collection forms, outcome measurement tools and the PERMIT intervention as a whole | 4 weeks
  The investigaotrs will use the weekly debrief with PERMIT champions, interviews with PICU health care professionals and interviews with parents/legal guardians to assess acceptability of all data collection forms, outcome measurement tools and the PERMIT intervention as a whole. These data, along with the data from the data collection forms and outcome measurement tools themselves, will also provide the investigaotrs with an indication of the potential impact of the PERMIT intervention on CYP and parents/legal guardians.
Number of ERM activities prescribed per CYP following patient acuity screening | 4 weeks
  The Local PERMIT Research Team will record the number of ERM activities prescribed to CYP follow daily acuity screening daily.
Number of ERM activities delivered per CYP | 4 weeks
  The Local PERMIT Research Team will convert prescribed ERM activity to delivered ERM activity and will calculate this on a daily basis.

CONTACTS AND LOCATIONS:
Overall Officials: Barnaby Scholefield, Dr, Study Chair — Birmingham Women's and Children's Hospital
Locations (1):
- Birmingham Women and Children's Hospital PICU, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Scholefield BR, Menzies JC, McAnuff J, Thompson JY, Manning JC, Feltbower RG, Geary M, Lockley S, Morris KP, Moore D, Pathan N, Kirkham F, Forsyth R, Rapley T. Implementing early rehabilitation and mobilisation for children in UK paediatric intensive care units: the PERMIT feasibility study. Health Technol Assess. 2023 Nov;27(27):1-155. doi: 10.3310/HYRW5688. PMID 38063184